CLINICAL TRIAL: NCT00063999
Title: Randomized Phase III Trial of Doxorubicin/Cisplatin/Paclitaxel and G-CSF Versus Carboplatin/Paclitaxel in Patients With Stage III &Amp; IV or Recurrent Endometrial Cancer
Brief Title: Doxorubicin Hydrochloride, Cisplatin, and Paclitaxel or Carboplatin and Paclitaxel in Treating Patients With Stage III-IV or Recurrent Endometrial Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GOG Foundation (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GOG-0209; NCI-2009-00584 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000305940; GOG-0209 (Other: NRG Oncology); GOG-0209 (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2003-07-08; First posted 2003-07-09 (Estimated); Results first posted 2018-04-23 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-09

CONDITIONS: Recurrent Uterine Corpus Carcinoma; Stage IIIA Uterine Corpus Cancer AJCC v7; Stage IIIB Uterine Corpus Cancer AJCC v7; Stage IIIC Uterine Corpus Cancer AJCC v7; Stage IVA Uterine Corpus Cancer AJCC v7; Stage IVB Uterine Corpus Cancer AJCC v7
MeSH Terms: interventions — Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Doxorubicin; Filgrastim; Granulocyte Colony-Stimulating Factor; Paclitaxel; Taxes; pegfilgrastim

ARMS (2):
- Arm I (doxorubicin hydrochloride, cisplatin, paclitaxel) (Active Comparator): Patients receive doxorubicin hydrochloride IV over approximately 15-30 minutes on day 1, cisplatin IV over 60-90 minutes on day 1, paclitaxel IV over 3 hours on day 2, and filgrastim SC on days 3-12 or pegfilgrastim SC on day 3. Treatment repeats every 21 days for 7 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cisplatin; Drug: Doxorubicin Hydrochloride; Biological: Filgrastim; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Biological: Pegfilgrastim; Other: Quality-of-Life Assessment
- Arm II (paclitaxel, carboplatin) (Experimental): Patients receive paclitaxel IV over 3 hours and carboplatin IV over 30-60 minutes on day 1. Treatment repeats every 21 days for 7 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
  Arms: Arm II (paclitaxel, carboplatin)
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
  Arms: Arm I (doxorubicin hydrochloride, cisplatin, paclitaxel)
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
  Arms: Arm I (doxorubicin hydrochloride, cisplatin, paclitaxel)
Biological: Filgrastim — Given SC
  Other Names: FILGRASTIM, LICENSE HOLDER UNSPECIFIED; G-CSF; Neupogen; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; rG-CSF; Tevagrastim
  Arms: Arm I (doxorubicin hydrochloride, cisplatin, paclitaxel)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Biological: Pegfilgrastim — Given SC
  Other Names: Filgrastim SD-01; filgrastim-SD/01; Fulphila; HSP-130; Jinyouli; Neulasta; Neulastim; Pegfilgrastim Biosimilar HSP-130; SD-01; SD-01 sustained duration G-CSF
  Arms: Arm I (doxorubicin hydrochloride, cisplatin, paclitaxel)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This randomized phase III trial compares how well two different combination chemotherapy regimens (doxorubicin hydrochloride, cisplatin, and paclitaxel versus carboplatin and paclitaxel) work in treating patients with endometrial cancer that is stage III-IV or has come back (recurrent). Drugs used in chemotherapy such as doxorubicin hydrochloride, cisplatin, paclitaxel, and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known which combination chemotherapy regimen is more effective in treating endometrial cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if the combination of carboplatin and paclitaxel (TC) chemotherapy is therapeutically equivalent to the combination of doxorubicin (doxorubicin hydrochloride), cisplatin and paclitaxel (TAP) chemotherapy with regards to survival.

II. To determine if estrogen/progesterone receptor status provides prognostic information in patients treated with chemotherapy.

III. To assess whether combination TC chemotherapy is superior to combination TAP chemotherapy with regards to toxicity profile, specifically neurotoxicity and infection.

IV. To measure differences in patient-reported neurotoxicity and quality of life (QOL) among the regimens.

OUTLINE: Patients are randomized to 1 of 2 treatment arms. Patients with left ventricular ejection fraction < 50% at randomization who are initially randomized to Arm I are immediately crossed over to Arm II.

ARM I: Patients receive doxorubicin hydrochloride intravenously (IV) over approximately 15-30 minutes on day 1, cisplatin IV over 60-90 minutes on day 1, paclitaxel IV over 3 hours on day 2, and filgrastim subcutaneously (SC) on days 3-12 or pegfilgrastim SC on day 3.

ARM II: Patients receive paclitaxel IV over 3 hours and carboplatin IV over 30-60 minutes on day 1.

In both arms, treatment repeats every 21 days for 7 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have primary stage III or stage IV or recurrent endometrial carcinoma whose potential for cure by radiation therapy or surgery alone or in combination is very poor; pathological confirmation and estrogen receptor (ER)/progesterone receptor (PR) status of the primary tumor is mandatory; however, the results do not need to be available prior to registration
* Patients may not have received prior cytotoxic chemotherapy, including chemotherapy used for radiation sensitization; patients may have received prior radiation therapy, hormonal therapy, or therapy with biologic agents, but such therapies must be discontinued prior to entry on this study
* Patients in whom both radiation and chemotherapy is planned must receive radiation prior to entry on this study; at least four weeks should have elapsed since completion of radiation therapy (RT) involving the whole pelvis or over 50% of the spine
* Platelets >= 100,000/mcl
* Granulocytes (absolute neutrophil count [ANC]) >= 1,500/mcl
* Creatinine =< upper limit of normal (ULN) (Common Toxicity Criteria [CTC] grade 0) or calculated creatinine clearance (Jeliffe Formula) >= 60 ml/min
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 3 x upper limits of normal
* Bilirubin =< institutional upper limits of normal
* Patients must have a Gynecologic Oncology Group (GOG) performance status of 0, 1, or 2
* Patients must have met the pre-entry requirements
* Patients must have signed an approved informed consent and authorization permitting release of personal health information

Exclusion Criteria:

* Patients with a concomitant malignancy other than non-melanoma skin cancer; with the exception of non-melanoma skin cancer, patients with a prior invasive malignancy who have been disease-free for < 5 years or who received prior chemotherapy for that malignancy
* Patients in whom pathological confirmation and estrogen receptor (ER)/progesterone receptor (PR) status of the tumor is not obtainable
* Patients for whom radiation therapy is planned during or after study chemotherapy prior to demonstrated progression
* Patients with concomitant medical illness such as serious uncontrolled infection, uncontrolled angina, or serious peripheral neuropathy, which, in the opinion of the treating physician, make the treatments prescribed on this study unreasonably hazardous for the patient
* Patients with third degree or complete heart block are not eligible unless a pacemaker is in place; patients on medications which alter cardiac conduction, such as digitalis, beta-blockers, or calcium channel blockers, or who have other conduction abnormalities or cardiac dysfunction may be placed on study at the discretion of the investigator
* Patients with history of myocardial infarct within 6 months before enrollment, New York Heart Association (NYHA) class II or greater heart failure or symptoms suspicious for congestive heart failure are not eligible unless a left ventricular ejection fraction in the past 6 months is documented to be 50% or greater; patients who have had a left ventricular ejection fraction (LVEF) (performed for any reason) of less than 50% in the past 6 months are ineligible
* Patients whose circumstances will not permit study completion or adequate follow-up
* Patients who are sensitive to E. coli-derived drug preparations
* Patients with uterine carcinosarcoma or other non-epithelial uterine malignancies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1381 (Actual)
Dates: Start 2003-08-25 (Actual); Primary Completion 2013-06-29 (Actual); Study Completion 2021-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David S Miller, Principal Investigator — NRG Oncology
Locations (650):
- United States (631):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Clearview Cancer Institute, Huntsville, Alabama
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Providence Hospital, Mobile, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Highlands Oncology Group PA - Fayetteville, Fayetteville, Arkansas
  - Washington Regional Medical Center - Fayetteville, Fayetteville, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - John Muir Medical Center-Concord Campus, Concord, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Saint Jude Medical Center, Fullerton, California
  - Marin Cancer Care Inc, Greenbrae, California
  - Long Beach Memorial Medical Center-Todd Cancer Institute, Long Beach, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Community Hospital of Los Gatos, Los Gatos, California
  - Doctors Medical Center, Modesto, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Oakland, Oakland, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - Salinas Valley Memorial, Salinas, California
  - University of California San Diego, San Diego, California
  - Alvarado Hospital Medical Center, San Diego, California
  - Zuckerberg San Francisco General Hospital, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Cancer Center of Santa Barbara, Santa Barbara, California
  - Ridley-Tree Cancer Center, Santa Barbara, California
  - Sansum Clinic Inc, Santa Barbara, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Ridley-Tree Cancer Center-Solvang, Solvang, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Olive View-University of California Los Angeles Medical Center, Sylmar, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - Colorado Gynecologic Oncology Group, Aurora, Colorado
  - University of Colorado, Denver, Colorado
  - Rocky Mountain Gynecologic Oncology PC, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Yale University, New Haven, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Saint Francis Hospital - Wilmington, Wilmington, Delaware
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Morton Plant Hospital, Clearwater, Florida
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Florida Gynecologic Oncology, Fort Myers, Florida
  - Saint Vincent's Medical Center, Jacksonville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - Mercy Hospital, Miami, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Bayfront Outpatient Health Clinic, St. Petersburg, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Florida Cancer Specialists-West Palm Beach, West Palm Beach, Florida
  - Southeastern Gynecologic Oncology LLP, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Atlanta Regional CCOP, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Dekalb Medical Center, Decatur, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Northside Hospital - Gwinnett, Lawrenceville, Georgia
  - Central Georgia Gynecologic Oncology, Macon, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Harbin Clinic Medical Oncology and Clinical Research, Rome, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Pacific Cancer Institute of Maui, Wailuku, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Anthony's Health, Alton, Illinois
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Rush - Copley Medical Center, Aurora, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Eureka Hospital, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Saint Francis Hospital, Evanston, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hinsdale Hematology Oncology Associates Incorporated, Hinsdale, Illinois
  - Hopedale Medical Complex - Hospital, Hopedale, Illinois
  - Duly Health and Care Joliet, Joliet, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Franciscan St. James Health-Olympia Fields Campus, Olympia Fields, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Chicago Gynecologic Oncology SC, Palatine, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - OSF Saint Anthony Medical Center, Rockford, Illinois
  - Sarah Culbertson Memorial Hospital, Rushville, Illinois
  - Saint Margaret's Hospital, Spring Valley, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Franciscan Saint Francis Health-Beech Grove, Beech Grove, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - McFarland Clinic PC - Ames, Ames, Iowa
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - Saint Luke's Hospital, Cedar Rapids, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Genesis Medical Center - East Campus, Davenport, Iowa
  - Genesis Cancer Care Institute, Davenport, Iowa
  - Mercy Capitol, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Providence Medical Center, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Radiation Oncology Practice Corporation Southwest, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Ascension Via Christi - Pittsburg, Pittsburg, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Advent Health - Shawnee Mission Medical Center, Shawnee Mission, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Saint Elizabeth Medical Center South, Edgewood, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Hospital Pavilion and Medical Campus, Louisville, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Woman's Hospital, Baton Rouge, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Maine Medical Center-Bramhall Campus, Portland, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - University of Maryland Shore Medical Center at Easton, Easton, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Kaiser Permanente - Largo Medical Center, Largo, Maryland
  - Kaiser Permanente - Towson Medical Center, Lutherville, Maryland
  - Kaiser Permanente - Shady Grove Medical Center, Rockville, Maryland
  - TidalHealth Peninsula Regional, Salisbury, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Dana Farber Community Cancer Care-Quincy, Quincy, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Beaumont Hospital - Dearborn, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Spectrum Health-Blodgett Campus, Grand Rapids, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Kalamazoo Center for Medical Studies, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Mercy Health Partners-Hackley Campus, Muskegon, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Ascension Providence Hospitals - Southfield, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Saint Dominic-Jackson Memorial Hospital, Jackson, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Keesler Medical Center, Keesler Air Force Base, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - Southeast Missouri Hospital, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Freeman Health System, Joplin, Missouri
  - Truman Medical Centers, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Radiation Oncology Practice Corporation South, Kansas City, Missouri
  - Saint Joseph Health Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Radiation Oncology Practice Corporation - North, Kansas City, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - SSM Health Saint Louis University Hospital, St Louis, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Saint Mary's Hospital, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Center for Cancer Care and Research, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Saint Louis-Cape Girardeau CCOP, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Deaconess Medical Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Internal Medicine of Bozeman, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Eastern Montana Cancer Center, Miles City, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Bryan LGH Medical Center West, Lincoln, Nebraska
  - Bryan LGH Medical Center East, Lincoln, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Center of Hope at Renown Medical Center, Reno, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Women's Cancer Center at Washoe, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Hunterdon Medical Center, Flemington, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Mountainside Hospital, Montclair, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Inspira Medical Center Mullica Hill, Mullica Hill, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - AtlantiCare Regional Medical Center -Main Campus, Pomona, New Jersey
  - Riverview Medical Center/Booker Cancer Center, Red Bank, New Jersey
  - Sparta Cancer Treatment Center, Sparta, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Southwest Gynecologic Oncology Associates Inc, Albuquerque, New Mexico
  - New York Oncology Hematology PC - Albany Medical Center, Albany, New York
  - Women's Cancer Care Associates LLC, Albany, New York
  - New York Oncology Hematology PC - Amsterdam, Amsterdam, New York
  - Island Gynecologic Oncology, Brightwaters, New York
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - New York Oncology Hematology PC - Clifton Park, Clifton Park, New York
  - New York Oncology Hematology PC-Hudson, Hudson, New York
  - Northwell Health NCORP, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - South Nassau Communities, Oceanside, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Wakefield Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Good Samaritan Hospital Medical Center, West Islip, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Hope Women's Cancer Centers-Asheville, Asheville, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Moorehead Memorial Hospital, Eden, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Gynecologic Oncology Network, Greenville, North Carolina
  - Vidant Medical Center, Greenville, North Carolina
  - Vidant Oncology-Kinston, Kinston, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Wilson Medical Center, Wilson, North Carolina
  - Novant Health Oncology Specialists, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - Cleveland Clinic Akron General, Akron, Ohio
  - Saint Elizabeth Boardman Hospital, Boardman, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Cleveland Clinic Mercy Hospital, Canton, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - North Coast Cancer Care-Clyde, Clyde, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Dayton Veterans Affairs Medical Center, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Hematology Oncology Center Incorporated, Elyria, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Fremont Memorial Hospital, Fremont, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Saint Luke's Hospital, Maumee, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - UH Seidman Cancer Center at Salem Regional Medical Center, Salem, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Joseph Warren Hospital, Warren, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Three Rivers Community Hospital, Grants Pass, Oregon
  - Asante Health System, Medford, Oregon
  - Providence Medford Medical Center, Medford, Oregon
  - Rogue Valley Medical Center, Medford, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Compass Oncology Rose Quarter, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Marion Community Hospital, Carbondale, Pennsylvania
  - Mercy Fitzgerald Hospital, Darby, Pennsylvania
  - Oncology Hematology Associates of Northern Pennsylvania, DuBois, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Drexel University School of Medicine, Philadelphia, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Jefferson Torresdale Hospital, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Einstein Medical Center Philadelphia, Philadelphia, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Mercy Hospital, Scranton, Pennsylvania
  - Hematology and Oncology Associates of North East Pennsylvania, Scranton, Pennsylvania
  - Moses Taylor Hospital, Scranton, Pennsylvania
  - Scranton Hematology Oncology, Scranton, Pennsylvania
  - Associates In Hematology Oncology PC-Upland, Upland, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Main Line Health NCORP, Wynnewood, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - University of South Carolina School of Medicine, Columbia, South Carolina
  - South Carolina Oncology Associates PA, Columbia, South Carolina
  - Black Hills Obstetrics and Gynecology, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Chattanooga's Program in Women's Oncology, Chattanooga, Tennessee
  - East Tennessee State University, Johnson City, Tennessee
  - Southeast Gynecologic Oncology Associates, Knoxville, Tennessee
  - East Tennessee Baptist Hospital-Mercy Health Partners, Knoxville, Tennessee
  - Knoxville Gynecologic Cancer Specialists PC, Knoxville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - Clements University Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Texas Tech University Health Sciences Center-Lubbock, Lubbock, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Cottonwood Hospital Medical Center, Murray, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Intermountain Health Care, Salt Lake City, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - Northern Virginia Pelvic Surgery Associates, Annandale, Virginia
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Danville Regional Medical Center, Danville, Virginia
  - Kaiser Permanente - Fair Oaks Medical Center, Fairfax, Virginia
  - Southside Community Hospital, Farmville, Virginia
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Peninsula Cancer Institute-Gloucester, Gloucester, Virginia
  - Virginia Oncology Associates-Hampton, Hampton, Virginia
  - Rappahannock General Hospital, Kilmarnock, Virginia
  - Peninsula Cancer Institute-Newport News, Newport News, Virginia
  - Bon Secours Mary Immaculate Hospital, Newport News, Virginia
  - Virginia Oncology Associates - Lake Wright, Norfolk, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - Richmond Radiation Oncology Center, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Roanoke, Virginia
  - Carilion Clinic Gynecological Oncology, Roanoke, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Peninsula Cancer Institute-Williamsburg, Williamsburg, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Saint Agnes Hospital/Agnesian Cancer Center, Fond du Lac, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Ascension Columbia Saint Mary's Hospital Ozaukee, Mequon, Wisconsin
  - Ascension Columbia Saint Mary's Hospital - Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Ascension All Saints Hospital, Racine, Wisconsin
  - Ascension Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic - Slinger, Slinger, Wisconsin
  - Ascension Saint Michael's Hospital, Stevens Point, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Welch Cancer Center, Sheridan, Wyoming
- Canada (4):
  - McGill University Health Centre at Royal Victoria Hospital, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec
  - Saint Mary's Hospital, Montreal, Quebec
  - CHU de Quebec-L'Hotel-Dieu de Quebec (HDQ), Québec, Quebec
- Japan (15):
  - Tohoku University School of Medicine, Sendai, Aoba-ku
  - Kure National Hospital, Kure, Hiroshima
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Iwate Medical University Hospital, Shiwa-gun, Iwate
  - Kagoshima City Hospital, Kagoshima, Kagoshima-ken
  - Jikei University Aoto Hospital, Katsushika-ku, Tokyo
  - Keio University, Shinjuku-ku, Tokyo
  - Hiroshima University Hospital, Hiroshima
  - National Hospital Organization-Kobe Medical Center, Kobe
  - Shikoku Cancer Center, Matsuyama
  - National Kyushu Cancer Center, Minamiku
  - Jikei University School of Medicine, Minato-ku, Tokyo
  - Saitama Medical University International Medical Center, Saitama
  - National Cancer Center Hospital, Tokyo
  - Tottori University, Tottori

REFERENCES:
- [Derived] Miller DS, Filiaci VL, Mannel RS, Cohn DE, Matsumoto T, Tewari KS, DiSilvestro P, Pearl ML, Argenta PA, Powell MA, Zweizig SL, Warshal DP, Hanjani P, Carney ME, Huang H, Cella D, Zaino R, Fleming GF. Carboplatin and Paclitaxel for Advanced Endometrial Cancer: Final Overall Survival and Adverse Event Analysis of a Phase III Trial (NRG Oncology/GOG0209). J Clin Oncol. 2020 Nov 20;38(33):3841-3850. doi: 10.1200/JCO.20.01076. Epub 2020 Sep 29. PMID 33078978

RESULTS

PARTICIPANT FLOW:
Recruitment Details: GOG 0209 accrued 1381 patients from August 2003 to April 2009. 1312 of these patients were eligible.
Groups:
- Doxorubicin, Cisplatin, Paclitaxel: Patients receive doxorubicin IV over approximately 15-30 minutes on day 1, cisplatin IV over 60-90 minutes on day 1, paclitaxel IV over 3 hours on day 2, and filgrastim SC on days 3-12 or pegfilgrastim SC on day 3. Treatment repeats every 21 days for 7 courses in the absence of disease progression or unacceptable toxicity.
- Paclitaxel, Carboplatin: Patients receive paclitaxel IV over 3 hours and carboplatin IV over 30-60 minutes on day 1. Treatment repeats every 21 days for 7 courses in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Doxorubicin, Cisplatin, Paclitaxel | Paclitaxel, Carboplatin
Started | 692 | 689
Completed | 647 | 665
Not Completed | 45 | 24
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Ineligible | 44 | 24

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Doxorubicin Hydrochloride, Cisplatin, Paclitaxel) | Arm II (Paclitaxel, Carboplatin) | Total
Number analyzed (Participants) | 647 | 665 | 1312
Age, Customized [Count of Participants; unit: Participants]
  <40 years | 19 | 18 | 37
  40 -49 years | 67 | 70 | 137
  50-59 years | 192 | 219 | 411
  60-60 years | 256 | 244 | 500
  >=70 years | 113 | 114 | 227
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 647 | 665 | 1312
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Alive at Time of Last Follow-up.
Description: The time alive in months from study entry to last contact or death.
Time Frame: Patients were assessed during treatment. Following completion of treatment, follow up was assessed every 3 months for 2 years, then every 6 months for 3 years and annually after for a maximum of 10 years.
Population: Eligible and treated patients. Data are reported from the second interim analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Arm I (Doxorubicin, Cisplatin, Paclitaxel): Patients receive doxorubicin IV over approximately 15-30 minutes on day 1, cisplatin IV over 60-90 minutes on day 1, paclitaxel IV over 3 hours on day 2, and filgrastim SC on days 3-12 or pegfilgrastim SC on day 3. Treatment repeats every 21 days for 7 courses in the absence of disease progression or unacceptable toxicity.
Arm/Group | Arm I (Doxorubicin, Cisplatin, Paclitaxel) | Arm II (Paclitaxel, Carboplatin)
Number analyzed (Participants) | 647 | 665
Participants
  Alive | 376 | 385
  Dead | 271 | 280

2. Secondary Outcome: Patient-reported Neurotoxicity (Ntx) as Measured by the FACT/GOG-Ntx Subscale (Short)
Description: The FACT/GOG-Ntx subscale (short version) contains 4 items measuring sensory neuropathy. Each item is scored using a 5-point Likert scale (0=not at all; 1= a little bit; 2=somewhat; 3=quite a bit; 4=very much). For east item, reversal was performed prior to score calculation so that a large score suggests less symptom. according to the FACIT measurement system, the subscale score was calculated as the summation of the individual item scores if more than 50% of subscale items were answered. When unanswered items existed, a subscale score was prorated by multiplying the mean of the answered item scores by the number of items in the subscale. The Ntx subscale score ranges 0-16 with a large subscale score suggests less symptom or better QOL (Quality of Life).
Time Frame: Baseline, 6 weeks post treatment start, 15 weeks post treatment start and 26 weeks post treatment start
Population: Eligible and evaluable and enrolled prior to 3/26/2006
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Doxorubicin, Cisplatin, Paclitaxel | Paclitaxel, Carboplatin
Number analyzed (Participants) | 228 | 246
units on a scale
  Baseline | 14.9 (0.15) | 14.9 (0.14)
  6 Weeks | 13.5 (0.28) | 11.3 (0.27)
  15 Weeks | 11.1 (0.37) | 11.2 (0.34)
  26 Weeks | 9.5 (0.41) | 10.9 (0.36)

3. Secondary Outcome: Patient Reported Quality of Life as Measured With the Combination of Physical Well-being (PWB) Subscale and Functional Well-being (FWB) Subscale From the FACT-G
Description: The FACT-G contains 4 subscales: Physical Well Being (7 items), Social Well Being (7 items), Emotional Well Being (6 items), Functional Well Being (7 items). The combination (14 items) of the physical well-being (PWB) and functional well-being (FWB) subscales was used to measure the HRQOL (Health Related Quality of Life). Each item is scored using a 5-point Likert scale (0=not at all; 1=a little bit; 2=somewhat; 3=quite a bit; 4=very much). for each negative item, reversal was performed prior to score calculation so that a large score suggests better QOL. A subscale score was calculated as the summation of the individual item scores if more than 50% of subscale items were answered. When unanswered items existed, a subscale score was prorated by multiplying the mean of the answred item scores by the number of items in the subscale. The QOL was measured with the summation of the PWB and FWBsubscale score and ranges 0-56 with a large score suggests better QOL.
Time Frame: Pre-treatment, 6 weeks post starting treatment (prior to cycle 3), 15 weeks post starting treatment (prior to cycle 6), 26 weeks post starting treatment
Population: Eligible and evaluable and enrolled prior to 3/26/2006
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Arm I (Doxorubicin, Cisplatin, Paclitaxel) | Arm II (Paclitaxel, Carboplatin)
Number analyzed (Participants) | 228 | 246
units on a scale
  Baseline | 39.4 (0.72) | 37.9 (0.7)
  6 weeks | 35.5 (0.73) | 37.5 (0.68)
  15 weeks | 35.3 (0.74) | 36.5 (0.7)
  26 weeks | 39.8 (0.8) | 38.5 (0.81)

4. Secondary Outcome: Number of Participants Alive at Time of Last Follow-up by Estrogen or Progesterone Receptor Status (Positive or Negative)
Description: The time alive in months from study entry to last contact or death.
Time Frame: Patients were assessed during treatment. Following completion of treatment, follow up was assessed every 3 months for 2 years, then every 6 months for 3 years and annually thereafter, for a maximum of 10 years.
Population: Eligible patients with estrogen and progesterone receptor data.
Measure: Count of Participants; unit: Participants
Groups:
- Estrogen Receptor Positive: Patients with estrogen receptor positive tumors
- Estrogen Receptor Negative: Patients with estrogen receptor negative tumors
- Progesterone Receptor Positive: Patients with progesterone receptor positive tumors
- Progesterone Receptor Negative: Patients with progesterone receptor negative tumors
Arm/Group | Estrogen Receptor Positive | Estrogen Receptor Negative | Progesterone Receptor Positive | Progesterone Receptor Negative
Number analyzed (Participants) | 919 | 355 | 832 | 440
Participants
  Alive | 408 | 90 | 380 | 117
  Dead | 511 | 265 | 452 | 323

5. Secondary Outcome: Number of Participants With Indicated Severity of CTCAE v2 Graded Neurotoxicity and Infection
Description: Maximum grade of physician assessed neurotoxicity and infection
Time Frame: Assessed throughout the treatment period and for 30 days after discontinuation of treatment.
Population: Eligible and treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Doxorubicin Hydrochloride, Cisplatin, Paclitaxel) | Arm II (Paclitaxel, Carboplatin)
Number analyzed (Participants) | 640 | 664
Participants
  Grade < 2 Sensory neuropathy | 167 | 130
  Grade 2 or Higher Sensory Neuropathy | 473 | 534
  Grade <3 infection with Neutrope | 25 | 29
  Grade 3 or Higher Infection with Neutropenia | 615 | 635
  Grade <3 infection without Neutropenia | 22 | 13
  Grade 3 or Higher Infection without Neutropenia | 618 | 651

ADVERSE EVENTS:
Time Frame: Adverse Events were recorded from the initiation of any study treatment up until 30 days following the last cycle of study treatment, up to 10 years.
Description: CTCAE v2.0 was used to grade and categorize all AEs and SAEs until 3/31/2010. Beginning 4/1/2010 CTCAE v4 was used to grade and categorize SAEs through AdEERs. All AEs and SAEs reported here were mapped to CTCAE v2.0.
Arm/Group | Arm I (Doxorubicin, Cisplatin, Paclitaxel) | Arm II (Paclitaxel, Carboplatin)
All-Cause Mortality (participants affected / at risk) | 271/647 | 280/665
Serious Adverse Events (participants affected / at risk) | 217/647 | 156/665
Other Adverse Events (participants affected / at risk) | 631/647 | 657/665
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Doxorubicin, Cisplatin, Paclitaxel) (N=647) | Arm II (Paclitaxel, Carboplatin) (N=665)
Allergic Reaction/Hypersensitivity (Immune system disorders) | 4 | 3
Hemoglobin (Blood and lymphatic system disorders) | 5 | 10
Hematologic-Other (Blood and lymphatic system disorders) | 0 | 1
Transfusion: Platelets (Blood and lymphatic system disorders) | 1 | 0
Transfusion: Prbcs (Blood and lymphatic system disorders) | 2 | 1
Platelets (Blood and lymphatic system disorders) | 4 | 5
Neutrophils/Granulocytes (Blood and lymphatic system disorders) | 16 | 26
Leukocytes (Blood and lymphatic system disorders) | 5 | 0
Hypertension (Cardiac disorders) | 1 | 0
Circulatory Or Cardiac-Other (Cardiac disorders) | 1 | 0
Cardiac Left Ventricular Function (Cardiac disorders) | 2 | 1
Hypotension (Cardiac disorders) | 0 | 2
Sinus Tachycardia (Cardiac disorders) | 1 | 0
Phlebitis (Cardiac disorders) | 1 | 0
Vasovagal Episode (Cardiac disorders) | 0 | 1
Supraventricular Arrhythmias (Cardiac disorders) | 2 | 1
Thrombosis/Embolism (Cardiac disorders) | 33 | 16
Cardiac-Ischemia/Infarction (Cardiac disorders) | 3 | 0
Sinus Bradycardia (Cardiac disorders) | 1 | 0
Prothrombin Time (Vascular disorders) | 1 | 0
Constitutional Symptoms-Other (General disorders) | 1 | 1
Fever In The Absence Of Neutropenia (General disorders) | 2 | 1
Fatigue (General disorders) | 5 | 1
Wound-Infectious (Skin and subcutaneous tissue disorders) | 2 | 3
Skin-Other (Skin and subcutaneous tissue disorders) | 1 | 0
Wound-Non-Infectious (Skin and subcutaneous tissue disorders) | 1 | 0
Stomatitis/Pharyngitis (Gastrointestinal disorders) | 1 | 0
Gi-Other (Gastrointestinal disorders) | 5 | 3
Fistula-Intestinal (Gastrointestinal disorders) | 1 | 1
Duodenal Ulcer (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 3 | 3
Gastritis (Gastrointestinal disorders) | 0 | 1
Mucositis Due To Radiation (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 2
Fistula-Rectal/Anal (Gastrointestinal disorders) | 1 | 1
Dehydration (Gastrointestinal disorders) | 16 | 9
Constipation (Gastrointestinal disorders) | 2 | 4
Diarrhea (Without Colostomy) (Gastrointestinal disorders) | 9 | 1
Vomiting (Gastrointestinal disorders) | 13 | 2
Nausea (Gastrointestinal disorders) | 7 | 3
Melena/Gi Bleeding (Vascular disorders) | 3 | 1
Vaginal Bleeding (Vascular disorders) | 2 | 1
Rectal Bleeding/Hematochezia (Vascular disorders) | 1 | 0
Hemorrhage/Bleeding Without Grade 3 Or 4 (Vascular disorders) | 1 | 0
Hepatic-Other (Hepatobiliary disorders) | 0 | 1
Sgot (Hepatobiliary disorders) | 1 | 1
Infection, Other (Infections and infestations) | 3 | 0
Catheter-Related Infection (Infections and infestations) | 6 | 1
Infection With Unknown Anc (Infections and infestations) | 1 | 1
Infection Documented W Grd 3/4 Neutropn. (Infections and infestations) | 18 | 9
Infection Without Neutropenia (Infections and infestations) | 17 | 8
Febrile Neutropenia-Fuo Infect Not Docum (Infections and infestations) | 14 | 14
Lymphatics-Other (Blood and lymphatic system disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 3 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 2
Hypokalemia (Metabolism and nutrition disorders) | 5 | 2
Hypomagnesmia (Metabolism and nutrition disorders) | 4 | 0
Muscle Weakness Not Due To Neuropathy (Musculoskeletal and connective tissue disorders) | 3 | 1
Tremor (Nervous system disorders) | 1 | 0
Neurologic-Other (Nervous system disorders) | 1 | 2
Seizure(S) (Nervous system disorders) | 1 | 0
Depressed Level Of Consciousness (Nervous system disorders) | 0 | 1
Cns Cerebrovascular Ischemia (Nervous system disorders) | 3 | 1
Confusion (Nervous system disorders) | 0 | 1
Ataxia (Nervous system disorders) | 0 | 2
Syncope (Nervous system disorders) | 1 | 1
Mood Alteration-Anxiety Agitation (Nervous system disorders) | 0 | 1
Mood Alteration-Depression (Nervous system disorders) | 3 | 0
Neuropathy-Sensory (Nervous system disorders) | 2 | 1
Neuropathy Motor (Nervous system disorders) | 0 | 2
Ocular-Other (Eye disorders) | 0 | 1
Chest Pain Non-Cardiac Or Non-Pleuritic (General disorders) | 1 | 4
Rectal Or Perirectal Pain (General disorders) | 0 | 1
Abdominal Pain Or Cramping (General disorders) | 6 | 4
Pain-Other (General disorders) | 0 | 1
Pneumonitis/Pulmonary Infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural Effusion (Non-Malignant) (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Pulmonary-Other (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Adult Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Ureteral Obstruction (Renal and urinary disorders) | 0 | 3
Fistula Or Gu Fistula (Renal and urinary disorders) | 0 | 1
Renal Failure (Renal and urinary disorders) | 0 | 1
Creatinine (Renal and urinary disorders) | 4 | 2
Renal/Gu-Other (Renal and urinary disorders) | 2 | 1
Syndromes-Other (General disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Doxorubicin, Cisplatin, Paclitaxel) (N=647) | Arm II (Paclitaxel, Carboplatin) (N=665)
Leukocytes (Blood and lymphatic system disorders) | 418 | 556
Neutrophils/Granulocytes (Blood and lymphatic system disorders) | 402 | 590
Platelets (Blood and lymphatic system disorders) | 244 | 172
Hemoglobin (Blood and lymphatic system disorders) | 445 | 410
Hematologic-Other (Blood and lymphatic system disorders) | 202 | 156
Allergic Reaction/Hypersensitivity (Immune system disorders) | 18 | 29
Ear and labyrinth disorders (Ear and labyrinth disorders) | 26 | 13
Cardiac Left Ventricular Function (Cardiac disorders) | 50 | 0
Cardiac disorders (Cardiac disorders) | 55 | 40
Vascular disorders (Vascular disorders) | 5 | 4
Constitutional (General disorders) | 37 | 26
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 473 | 486
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 25 | 12
Endocrine disorders (Endocrine disorders) | 11 | 7
All other GI (Gastrointestinal disorders) | 163 | 125
Nausea (Gastrointestinal disorders) | 218 | 122
Vomiting (Gastrointestinal disorders) | 165 | 82
Stomatitis/Pharyngitis (Gastrointestinal disorders) | 54 | 17
Renal and urinary disorders (Renal and urinary disorders) | 15 | 20
Vascular disorders (Vascular disorders) | 6 | 7
Hepatobiliary disorders (Hepatobiliary disorders) | 17 | 17
Infections and infestations (Infections and infestations) | 19 | 8
Febrile Neutropenia-Fuo Infect Not Docum (Infections and infestations) | 45 | 37
Infection Without Neutropenia (Infections and infestations) | 54 | 25
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 7 | 3
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 140 | 96
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 24 | 20
Nervous system disorders (Nervous system disorders) | 67 | 47
Neuropathy: sensory (Nervous system disorders) | 163 | 128
Eye disorders (Eye disorders) | 46 | 34
Pain (General disorders) | 91 | 89
myalgia (General disorders) | 95 | 97
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 90 | 82
Neoplasms benign, malignant and unspecified (including cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3

LIMITATIONS AND CAVEATS:
Eligibility for this study was expanded from measurable, stage 3 or stage 4 or recurrent disease to include non-measurable, stage 4 or recurrent disease and then to include non-measurable stage 3 disease.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less